CLINICAL TRIAL: NCT01408238
Title: Biological Standardization of Secale Cereale Allergen Extract to Determine the Biological Activity in Histamine Equivalent Prick (HEP) Units
Brief Title: Biological Standardization of Secale Cereale Allergen Extract
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laboratorios Leti, S.L. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 6049-PR-PRI-184; 2010-023951-27 (EudraCT Number)
Record Dates: First submitted 2011-08-01; First posted 2011-08-03 (Estimated); Last update posted 2012-08-09 (Estimated); Status verified 2012-08

CONDITIONS: Allergy to Grass Pollen (Secale Cereale)
Keywords: Immunotherapy; Skin prick test; Standardization; Secale cereale

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): * Secale cereale allergen extract at 4 different concentrations
  * Positive control
  * Negative control
  Interventions: Biological: Four different concentrations of Secale cereale allergen extract, positive control and negative control

INTERVENTIONS:
Biological: Four different concentrations of Secale cereale allergen extract, positive control and negative control — 4 concentrations of Secale cereale allergen extract, together with a positive and negative control will be tested in every patient in duplicate on the volar surface of the forearm

SUMMARY:
The objective of this study is to determine the biologic activity of a Secale cereale allergen extract in histamine equivalent prick (HEP) units, in order to be used as in-house reference preparation (IHRP).

DETAILED DESCRIPTION:
This is an open, unblinded and non-randomized biological assay. The study design is a slight modification of the recommendations proposed by the Nordic Guidelines.

Four concentrations of Secale cereale allergen extract, together with a positive and negative control, using 10 mg/ml histamine dihydrochloride solution and a glycerinated phenol saline solution, respectively, will be tested in every patient in duplicate on the volar surface of the forearm.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided written informed consent, appropriately signed and dated by the subject (or legal representative, if applicable).
2. Subject can be male or female of any race and ethnic group.
3. Age > 18 years and < 50 years at the study inclusion day.
4. Positive skin prick test with a standardized commercially available preparation of Secale cereale allergen extract. The skin prick test will be considered positive if the test results in a wheal major diameter of at least 3 mm and at least the size of the positive control. Positive skin prick test results are valid if performed within one year prior to the inclusion of the subject in the study
5. A positive test for specific IgE to Secale cereale (CAP-RAST ≥ 2). IgE results are valid if performed within one year prior to the inclusion of the subject in the study.
6. Allergic symptoms during the pollen season of Secale cereale.
7. Mean of the forearm major diameters of the wheals provoked by histamine dihydrochloride (10 mg/ml) ≥ 3 mm.

Exclusion Criteria:

1. Immunotherapy in the past 5 years with an allergen preparation known to interfere with the allergen to be tested (e.g., grass group extracts).
2. Use of drugs that may interfere with the skin reactions (e.g., antihistamines). See Appendix 1
3. Treatment with any of the following medications: tricyclic or tetracyclic antidepressants, β-blockers or corticosteroids (> 10 mg/day of prednisone or equivalent).
4. Pregnancy.
5. Dermographism affecting the skin area at the test site at either study visit.
6. Atopic dermatitis affecting the skin area at the test site at either study visit.
7. Urticaria affecting the skin area at the test site at either study visit.
8. Participation in another clinical trial within the last month.
9. Subjects suffering from pathologies or conditions in which adrenalin is contraindicated (heart disease, severe hypertension, ..)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2011-10; Primary Completion 2012-03 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Wheal size area (mm2) on the skin at the site of the puncture during the immediate phase. | Test sites should be inspected and recorded 15-20 min after application

CONTACTS AND LOCATIONS:
Overall Officials: María José Gómez, Study Chair — Laboratorios LETI, S.L.Unipersonal
Locations (2):
- Spain (2):
  - Hospital Universitario La Paz, Madrid, Madrid / Madrid
  - Hospital Universitario Virgen Macarena, Seville, Sevilla / Andalucía